CLINICAL TRIAL: NCT02803970
Title: Establishing the Registry of Korean Patients With Borderline Ovarian Tumors
Brief Title: KOrean Borderline Ovarian Tumor (KOBOT) Registry
Acronym: KOBOT
Status: Recruiting | Type: Observational
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Other Study IDs: 2015-08-002
Record Dates: First submitted 2016-06-11; First posted 2016-06-17 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to collect data on Korean patients with borderline ovarian tumors.

DETAILED DESCRIPTION:
The researchers retrospectively collected data on Korean patients with borderline ovarian tumors (BOTs) diagnosed, treated, and followed between November 1994 and February 2015 at institutions where placed in the Republic of Korea. And the researchers prospectively will collect data on all Korean patients with BOTs at institutions where placed in the Republic of Korea since March, 2015. If patients agree to participate in this KOBOT registry, patient's data (such as age, body mass index, preoperative findings, laboratory findings, radiologic findings, operative findings, pathologic findings, postoperative findings) will be collected in a research database. The research database will be updated, every 6 month, to include data on patient's disease outcome and follow-up care. Although most data will be collected form the medical record, patient may agin be contacted so that researchers can collection some data if it is not in the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patients with borderline ovarian tumors (BOTs) diagnosed, treated, and followed between November 1994 and February 2015 at institutions where placed in the Republic of Korea.
* All patients undergoing gynecologic surgery for BOTs at institutions where placed in the Republic of Korea since March, 2015

Exclusion Criteria:

* Patients who did not receive primary treatment or follow-up for at least 6 months at each institution were excluded from analysis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean patients with borderline ovarian tumors (BOTs)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 1994-12; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD, PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (4):
- South Korea (4):
  - Samsung Changwon Hospital, Changwon
  - Kangbuk Samsung Hospital, Seoul
  - CHA Gangnam Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No